CLINICAL TRIAL: NCT03905239
Title: Impact of a Procalcitonin-based Algorithm on Quality of Management in Patients With Uncomplicated Adhesion-related Small Bowel Obstruction Assessed by Textbook Outcome: a Multicenter Cluster-randomized Open-label Controlled Trial. (ALPROC)
Brief Title: A Procalcitonin-based Algorithm in Adhesion-related Small Bowel Obstruction
Acronym: ALPROC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Centre Hospitalier de Beauvais (Other); University Hospital, Rouen (Other); University Hospital, Caen (Other); University Hospital, Lille (Other); Groupe Hospitalier Pitie-Salpetriere (Other); Centre Hospitalier Universitaire Dijon (Other); University Hospital, Limoges (Other); Saint Antoine University Hospital (Other); University Hospital, Clermont-Ferrand (Other); Hôpital Cochin (Other); University Hospital, Toulouse (Other); Centre Hospitalier de PAU (Other); Hopital Lariboisière (Other); Tourcoing Hospital (Other); Central Hospital Saint Quentin (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PI2018_843_0029
Record Dates: First submitted 2019-02-21; First posted 2019-04-05 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Small Bowel Obstruction
Keywords: algorithm; procalcitonin; small bowel obstruction
MeSH Terms: interventions — Algorithms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- algorithm arm (Experimental): Patient management is based on clinical examination and procalcitonin assessment. From 48 hours after initiation of conservative management in the case of absence of bowel function, operative management (adhesiolysis or bowel resection) will be performed. In the event of discordance between procalcitonin values and clinical examination, management will always be based on clinical examination.
  Interventions: Diagnostic Test: algorithm
- no algorithm arm (No Intervention): Patient management is based on clinical examination. Conservative management will be continued for 48 hours in the absence of signs of bowel ischemia (clinical and laboratory assessment other than procalcitonin, as procalcitonin will not be assayed in this arm). Gastrografin will not be used in this arm. Operative management (adhesiolysis or bowel resection) will be performed 48 hours after initiation of conservative management or in the case of absence of bowel function.

INTERVENTIONS:
Diagnostic Test: algorithm — clinical examination and procalcitonin assessment
  Arms: algorithm arm

SUMMARY:
Adhesion-related small bowel obstruction is a common digestive emergency that can be managed either conservatively or surgically. However, the choice between these two approaches can be difficult due to the absence of specific signs. The objective of this study is to evaluate the clinical impact of a procalcitonin-based algorithm.

DETAILED DESCRIPTION:
Acute adhesion-related small bowel obstruction (ASBO) is a common digestive emergency accounting for 1% to 3% of all digestive emergencies. It is associated with a mortality rate of between 2% and 8%, although this figure may be as high as 25% when surgical treatment is delayed. In 2013, the World Society of Emergency Surgery's working group on ASBO suggested two distinct approaches for the management of acute ASBO. Conservative management includes the use of a nasogastric tube (NGT), intravenous administration of fluids, and clinical and biochemical monitoring for 24 to 72 hours or surgical management. However, the efficacy of conservative management in this setting is a subject of debate, as it might delay the decision to perform surgery and increase the frequency of bowel resection (e.g. in the presence of bowel necrosis) or, in contrast, prompt an excessive number of unnecessary laparotomies. The efficacy of water-soluble contrast medium in this setting is also subject to debate, as data from a recent randomized clinical trial including 242 patients (ABOD study) combined with a meta-analysis in 2015 including 990 patients failed to demonstrate any value of gastrografin to reduce the surgery rate and length of stay. Three years ago, our team proposed the use of a marker of bacterial infection and bowel ischemia, procalcitonin (PCT), to help distinguish patients in whom conservative management is likely to be successful from those in whom surgical management was mandatory. Cutoffs of 0.2 µg/L (for failure of conservative management ) and 0.6 µg/L (for need for surgery) accurately identified more than 80% of patients. These cutoffs and data were confirmed in a second independent cohort, and were then used to propose an algorithm for the management of patients with ASBO. In this single-center, retrospective , case-control study, the investigators showed that introduction of this algorithm into patient management reduced i/ the time to surgery with no increase of the surgical management rate; ii/ the length of stay (with a 2-day difference). The investigators propose the hypothesis that introduction of the PCT-based algorithm improves the quality of management of patients with ASBO.

ELIGIBILITY:
Inclusion Criteria:

* Uncomplicated acute adhesion-related small bowel obstruction (ASBO)
* Adults
* Patients able to express consent
* Signed written informed consent form
* Covered by national health insurance

Exclusion Criteria:

* Disease-related criteria:
* Large bowel obstruction
* No previous abdominal surgery
* Signs of peritonitis or strangulation requiring emergency surgery)
* Obstruction within 4 weeks following previous surgery
* Ongoing or history of bowel cancer
* Ongoing or in history of inflammatory bowel disease
* History of abdominal radiotherapy
* Active infection
* Contraindication to contrast-enhanced CT scan
* Minors
* Patient deprived of liberty by administrative or judicial decision or placed under judicial protection (guardianship or supervision)
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
proportion of patients achieving textbook outcome | within 90 days after randomization.
  textbook outcome is defined as patients either correctly operated (ischemia confirmed at operation ± resection) or correctly managed conservatively (no need for unplanned surgery) with no major postoperative complications (Clavien-Dindo≥3) and a medical length of stay<5 days (defined as the time at which the patient is medically eligible for discharge), with no postoperative consultation, rehospitalisation and reoperation within 90 days after randomization.

SECONDARY OUTCOMES:
1-, 3-, 6-, 9-, 12-month recurrence rates | within 12 postoperative months
  a new episode of adhesion-related small bowel obstruction.
QSH45 (questionnaire for satisfaction of hospitalized patients) score evaluating patient satisfaction at postoperative month 1 | postoperative month 1
  Evaluation of patient satisfaction at postoperative month 1. Values of scores are between 0 and 100. 0 is the minimum score. 100 is the maximum score. In QSH45 : 45 questions are asked to the patient. Each question has a score from 1 (worst) to 5 (best score). The QSH45 score is divided in 8 subscales. The 45 questions are placed equally in the 8 subscales. the total score (QSH45) is the average of the score of the 8 subscales.
Clavien score postoperative month 1 | postoperative month 1
  The therapy used to correct a specific complication in the basis of this classification on order to rank a complication in an objective and reproducible manner. It consists of 7 grades (I, II, IIIa, IIIb, IVa, IVb and V). Grade I is the minimum value of the score. Grade V is the maximum value of the score corresponding to the death of a patient.
CCI score | postoperative month 1
  The CCI calculator is an online tool to support the assessment of patients' overall morbidity. The comprehensive complication index (CCI) is based on the complication grading by Clavien-Dindo Classification and implements every occured complication after an intervention. The overall morbidity is reflected on a scale from 0 (no complication) to 100 (death).
Hospital length of stay | postoperative month 12
  the interval between admission to the emergency department and discharge from the ward.
Cumulative length of stay | postoperative month 12
  total number of days of hospitalization related to ASBO

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc Regimbeau, Pr, Principal Investigator — CHU Amiens
Locations (1):
- Amiens Universitary Hospital, Amiens, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sabbagh C, Mauvais F, Tuech JJ, Tresallet C, Ortega-Debalon P, Mathonnet M, Lefevre JH, Lakkis Z, Fuks D, Muscari F, Dron B, Couderc P, Alves A, Regimbeau JM. Impact of a procalcitonin-based algorithm on the quality of management of patients with uncomplicated adhesion-related small bowel obstruction assessed by a textbook outcome: a multicenter cluster-randomized open-label controlled trial. BMC Gastroenterol. 2022 Mar 2;22(1):90. doi: 10.1186/s12876-022-02144-w. PMID 35236281